CLINICAL TRIAL: NCT06345118
Title: Evaluate the Results of Fall Prevention in Older Adults With Type 2 Diabetes Mellitus
Acronym: FallT2DMOLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Geriatric Hospital (Other Government)
Responsible Party: Principal Investigator, Dinh Trung Hoa, Endocrinologist Principal Investigator and Sponsor, National Geriatric Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FallpreventT2DMelderly
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Fall; Elderly Patient
Keywords: Falls prevention; Diabetes Mellitus type2; Elderly patient
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group receives supervised Otago exercise program and baseline treatment for type2 diabetes mellitus:
  The Otago exercise program aims to increase muscle strength and improve the patient's balance. The training duration is 24 weeks, the frequency is thrice a week, and the intensity gradually increases based on the Personal Therapist (PT) assessment.
  Baseline treatment for diabetes: Recommendations according to American Diabetes Association guidelines, which include instructions to follow the diet and exercises as recommended for older type 2 diabetic patients
  Interventions: Behavioral: Otago exercise program
- Control group (No Intervention): The control group receives the baseline treatment for type2 diabetes mellitus:
  Baseline treatment for diabetes: Recommendations according to American Diabetes Association guidelines, which include instructions to follow the diet and exercises as recommended for older type 2 diabetic patients

INTERVENTIONS:
Behavioral: Otago exercise program — The OEP consists of 17 strength and balance exercises and a walking program performed thrice a week by the older adult at home.
  Program Prescription The program is designed to be delivered over 6 months and includes a minimum of 5 visits. The first visit is Day 1 of Otago when performance of the functional measures is assessed, and the exercises are prescribed at the Rehabilitation Center of the National Geriatric Hospital. Then, the therapist will see the patient for 4 visits over an 8-week period (typically every other week). This is considered the initial bolus of Otago. Then, the therapist will follow the patient via phone calls every week and make a visit at three months, four months, five months, and six months to reassess the patient's training ability and compliance.
  Monitoring:
  Calendars can be completed each month to document any falls. A calendar or diary can be used to monitor compliance with the exercise programme
  Other Names: OEP
  Arms: Intervention group

SUMMARY:
.This randomized controlled clinical trial aims to evaluate the effects of fall prevention in older adults with type 2 diabetes mellitus. The main questions it aims to answer are:

* Describe the current situation of falls, the risk of falls, and some related factors in elderly type 2 diabetic patients
* Evaluate the results of fall prevention and related factors in the study population.

Participants will be randomly divided into control and intervention groups. The intervention group will be trained to follow the Otago Training Program as the primary fall prevention method. On the other hand, the control group will receive the standard care following the treatment guidelines for type 2 diabetes mellitus and other comorbidities.

At the end of the intervention, the study will mainly compare the rate of fall incidents after 6 months of intervention as well as other physical performance tests.

DETAILED DESCRIPTION:
The proportion of the elderly population is increasing remarkably worldwide. The United Nations estimates there will be 727 million people aged 65 and older in 2020. According to the World Bank, Vietnam is one of the countries with the fastest population aging rate. Diabetes mellitus type 2 (T2DM) is a major public health problem, and the prevalence of T2DM increases exponentially with age. T2DM is also common in older people, and it has been estimated that approximately 25% of the patients with diabetes are over 65. There are an estimated 3.99 million people with diabetes aged 20-79 in 2021 in Vietnam, and this population will reach 6.01 million by 2045. Besides T2DM, the older adult is often faced with a myriad of health-related issues and problems, with falling being one primary concern for persons over 65 years of age. The high prevalence of falls in elderly individuals with DM is well established, with reported annual incidence rates up to 39%. Falls are linked to increased fracture risk and hospitalization for trauma. Recurrent falls can have a significant impact on social and physical activities, as well as quality of life. Falls cause about 2.8 million injuries treated in emergency departments annually, including over 800,000 hospitalizations and over 27,000 deaths. The entire cost of fall injuries in 2013 was $34 billion. The key to fall prevention is identifying persons at risk and implementing the appropriate intervention. Although there are standard fall prevention guidelines worldwide, such as those of the American Geriatrics Society or the British Geriatrics Society, in Vietnam, there are no specific guidelines for screening and preventing falls for older people. Besides, the lack of research on the rate of falls in older people in Vietnam creates a gap in optimizing treatment for elderly diabetes patients, especially when diabetes complications are one of the leading causes of increased fall rates. This study aims to evaluate the rate of falls in elderly diabetic patients treated as outpatients at a National Geriatric Hospital (NGH) and then conduct fall prevention interventions using the Otago Exercise Program (OEP) as the primary method. The study will be submitted and approved by the National Geriatric Hospital Ethics Committee and Hanoi Medical University Ethics Committee, Vietnam, and written consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

For the first objective (Cross-sectional study):

* Type 2 diabetic patients diagnosed using American Diabetes Association 2022 criteria
* HbA1c ≥ 7.0 and ≤ 9%
* Age ≥ 60 and ≤ 80

For the second objective (Longitudinal study):

* All patients recruited from the first objective are at moderate or high risk of falls according to the criteria of World Guidelines for Falls Prevention and Management for Older Adults - British Geriatric Society.

Exclusion Criteria:

* Acute diabetic complications
* Patients are in the acute phase of musculoskeletal disorders: acute gout, progressing low-grade arthritis, acute joint pain due to joint degeneration, sciatic pain, and infectious arthritis.
* Patients suffer from conditions significantly affecting cognition and mobility: sequelae of stroke (with weakness, limb paralysis), muscular weakness, limb disabilities, severe heart failure, severe cognitive decline, and psychiatric disorders.
* Patients have been bedridden due to illness for more than one month within the past three months up to the recruitment time.
* Patients with cardiovascular diseases: chest pain, uncontrolled blood pressure ≥160/100 mmHg, untreated cardiac arrhythmia, a history of congestive heart failure, severe valvular heart disease, myocarditis or pericarditis, and hypertrophic cardiomyopathy.

Ages: 60 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical performance 1 - Timed Up and Go (TUG) | Prior to the start of intervention, reassess monthly at follow-up visits (1,2,3,4,5 month and 6th month - completion of intervention)
  To determine fall risk and measure the progress of balance, sit to stand and walking. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. Each group of patients will have different cut-off time value based on different studies
Physical performance 2 -Berg Balance Scale (BBS) | Prior to the start of intervention, reassess monthly at follow-up visits (1,2,3,4,5 month and 6th month - completion of intervention)
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. Cut-off scores for the elderly were reported by Berg et al 1992:
  A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling. A score of ≤49 indicates a risk of falls in individuals with stroke

SECONDARY OUTCOMES:
Activities of Daily Living (ADLs) | Prior to the start of intervention (Week 0), following the completion of the intervention (Week 24)
  Katz Index of Independence in Activities of Daily Living (scores range from 0-worst to 6-best)
Health-related Quality of Life | Prior to the start of intervention (Week 0), following the completion of the intervention (Week 24)
  Health-related Quality of Life is assessed using the health questionnaire 5-level 5 dimensions from EuroQol Group: index scores range from -0.59 to 1; 1 is the best possible health state.
Functional Reach Test (FRT) | Prior to the start of intervention, reassess monthly at follow-up visits (1,2,3,4,5 month and 6th month - completion of intervention)
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in in simple task.
  In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.
  This information is correlated with risk of falling. Measurement Interpretation: 10"/25 cm or greater: Low risk of falls; 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal; 6"/15cm or less Risk of falling is 4x greater than normal; Unwilling to reach: Risk of falling is 8x greater than normal
Instrumental Activities of Daily Living (IADLs) | Prior to the start of intervention (Week 0), following the completion of the intervention (Week 24)
  Lawton Instrumental Activities of Daily Living Scale (scores range from 0-low function & dependent to 8-high function & independent for women, and 0-worst to 5-best for men)

CONTACTS AND LOCATIONS:
Overall Officials: Huyen TT Vu, PhD, Study Chair — National Geriatric Hospital
Locations (1):
- National Geriatric Hospital, Hanoi, Vietnam

REFERENCES:
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S64-71. doi: 10.2337/dc12-s064. No abstract available. PMID 22187472
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] Montero-Odasso MM, Kamkar N, Pieruccini-Faria F, Osman A, Sarquis-Adamson Y, Close J, Hogan DB, Hunter SW, Kenny RA, Lipsitz LA, Lord SR, Madden KM, Petrovic M, Ryg J, Speechley M, Sultana M, Tan MP, van der Velde N, Verghese J, Masud T; Task Force on Global Guidelines for Falls in Older Adults. Evaluation of Clinical Practice Guidelines on Fall Prevention and Management for Older Adults: A Systematic Review. JAMA Netw Open. 2021 Dec 1;4(12):e2138911. doi: 10.1001/jamanetworkopen.2021.38911. PMID 34910151
- [Background] 2019 surveillance of falls in older people: assessing risk and prevention (NICE guideline CG161) [Internet]. London: National Institute for Health and Care Excellence (NICE); 2019 May 23. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK551819/ PMID 31869045
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Lee PG, Halter JB. The Pathophysiology of Hyperglycemia in Older Adults: Clinical Considerations. Diabetes Care. 2017 Apr;40(4):444-452. doi: 10.2337/dc16-1732. PMID 28325795
- [Background] Chia CW, Egan JM, Ferrucci L. Age-Related Changes in Glucose Metabolism, Hyperglycemia, and Cardiovascular Risk. Circ Res. 2018 Sep 14;123(7):886-904. doi: 10.1161/CIRCRESAHA.118.312806. PMID 30355075
- [Background] American Diabetes Association Professional Practice Committee. 13. Older Adults: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S195-S207. doi: 10.2337/dc22-S013. PMID 34964847
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S73-S84. doi: 10.2337/dc21-S006. PMID 33298417
- [Background] Kosorok MR, Omenn GS, Diehr P, Koepsell TD, Patrick DL. Restricted activity days among older adults. Am J Public Health. 1992 Sep;82(9):1263-7. doi: 10.2105/ajph.82.9.1263. PMID 1503169
- [Background] Scaf-Klomp W, van Sonderen E, Sanderman R, Ormel J, Kempen GI. Recovery of physical function after limb injuries in independent older people living at home. Age Ageing. 2001 May;30(3):213-9. doi: 10.1093/ageing/30.3.213. PMID 11443022
- [Background] McInnes L, Gibbons E, Chandler-Oatts J. Clinical practice guideline for the assessment and prevention of falls in older people. Worldviews Evid Based Nurs. 2005;2(1):33-6. doi: 10.1111/j.1524-475X.2005.04094.x. No abstract available. PMID 17040554
- [Background] Ortega-Bastidas P, Gomez B, Aqueveque P, Luarte-Martinez S, Cano-de-la-Cuerda R. Instrumented Timed Up and Go Test (iTUG)-More Than Assessing Time to Predict Falls: A Systematic Review. Sensors (Basel). 2023 Mar 24;23(7):3426. doi: 10.3390/s23073426. PMID 37050485
- [Background] Williams B, Allen B, Hu Z, True H, Cho J, Harris A, Fell N, Sartipi M. Real-Time Fall Risk Assessment Using Functional Reach Test. Int J Telemed Appl. 2017;2017:2042974. doi: 10.1155/2017/2042974. Epub 2017 Jan 10. PMID 28167961
- [Background] Greenberg SA. How to try this: the Geriatric Depression Scale: Short Form. Am J Nurs. 2007 Oct;107(10):60-9; quiz 69-70. doi: 10.1097/01.NAJ.0000292204.52313.f3. PMID 17895733
- [Background] Gregg EW, Beckles GL, Williamson DF, Leveille SG, Langlois JA, Engelgau MM, Narayan KM. Diabetes and physical disability among older U.S. adults. Diabetes Care. 2000 Sep;23(9):1272-7. doi: 10.2337/diacare.23.9.1272. PMID 10977018
- [Background] Yang Y, Hu X, Zhang Q, Zou R. Diabetes mellitus and risk of falls in older adults: a systematic review and meta-analysis. Age Ageing. 2016 Nov;45(6):761-767. doi: 10.1093/ageing/afw140. Epub 2016 Aug 11. PMID 27515679
- [Background] Sun J, Wang Y, Zhang X, Zhu S, He H. Prevalence of peripheral neuropathy in patients with diabetes: A systematic review and meta-analysis. Prim Care Diabetes. 2020 Oct;14(5):435-444. doi: 10.1016/j.pcd.2019.12.005. Epub 2020 Jan 6. PMID 31917119
- [Background] Najafi B, Horn D, Marclay S, Crews RT, Wu S, Wrobel JS. Assessing postural control and postural control strategy in diabetes patients using innovative and wearable technology. J Diabetes Sci Technol. 2010 Jul 1;4(4):780-91. doi: 10.1177/193229681000400403. PMID 20663438
- [Background] Lin SI, Chen YR, Liao CF, Chou CW. Association between sensorimotor function and forward reach in patients with diabetes. Gait Posture. 2010 Oct;32(4):581-5. doi: 10.1016/j.gaitpost.2010.08.006. Epub 2010 Sep 9. PMID 20829047
- [Background] Horak FB. Postural orientation and equilibrium: what do we need to know about neural control of balance to prevent falls? Age Ageing. 2006 Sep;35 Suppl 2:ii7-ii11. doi: 10.1093/ageing/afl077. PMID 16926210
- [Background] Morrison S, Colberg SR, Parson HK, Vinik AI. Relation between risk of falling and postural sway complexity in diabetes. Gait Posture. 2012 Apr;35(4):662-8. doi: 10.1016/j.gaitpost.2011.12.021. Epub 2012 Jan 23. PMID 22269128
- [Background] Haviv F, Ratajczyk JD, DeNet RW, Martin YC, Dyer RD, Carter GW. Structural requirements for the inhibition of 5-lipoxygenase by 15-hydroxyeicosa-5,8,11,13-tetraenoic acid analogues. J Med Chem. 1987 Feb;30(2):254-63. doi: 10.1021/jm00385a005. PMID 3806609
- [Background] van Dijk PT, Meulenberg OG, van de Sande HJ, Habbema JD. Falls in dementia patients. Gerontologist. 1993 Apr;33(2):200-4. doi: 10.1093/geront/33.2.200. PMID 8468012
- [Background] Coppin AK, Shumway-Cook A, Saczynski JS, Patel KV, Ble A, Ferrucci L, Guralnik JM. Association of executive function and performance of dual-task physical tests among older adults: analyses from the InChianti study. Age Ageing. 2006 Nov;35(6):619-24. doi: 10.1093/ageing/afl107. PMID 17047008
- [Background] Hausdorff JM, Yogev G, Springer S, Simon ES, Giladi N. Walking is more like catching than tapping: gait in the elderly as a complex cognitive task. Exp Brain Res. 2005 Aug;164(4):541-8. doi: 10.1007/s00221-005-2280-3. Epub 2005 Apr 28. PMID 15864565
- [Background] Chiu HL, Yeh TT, Lo YT, Liang PJ, Lee SC. The effects of the Otago Exercise Programme on actual and perceived balance in older adults: A meta-analysis. PLoS One. 2021 Aug 6;16(8):e0255780. doi: 10.1371/journal.pone.0255780. eCollection 2021. PMID 34358276
- [Result] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977
- [Result] Ganz DA, Latham NK. Prevention of Falls in Community-Dwelling Older Adults. N Engl J Med. 2020 Feb 20;382(8):734-743. doi: 10.1056/NEJMcp1903252. No abstract available. PMID 32074420
- [Result] James SL, Lucchesi LR, Bisignano C, Castle CD, Dingels ZV, Fox JT, Hamilton EB, Henry NJ, Krohn KJ, Liu Z, McCracken D, Nixon MR, Roberts NLS, Sylte DO, Adsuar JC, Arora A, Briggs AM, Collado-Mateo D, Cooper C, Dandona L, Dandona R, Ellingsen CL, Fereshtehnejad SM, Gill TK, Haagsma JA, Hendrie D, Jurisson M, Kumar GA, Lopez AD, Miazgowski T, Miller TR, Mini GK, Mirrakhimov EM, Mohamadi E, Olivares PR, Rahim F, Riera LS, Villafaina S, Yano Y, Hay SI, Lim SS, Mokdad AH, Naghavi M, Murray CJL. The global burden of falls: global, regional and national estimates of morbidity and mortality from the Global Burden of Disease Study 2017. Inj Prev. 2020 Oct;26(Supp 1):i3-i11. doi: 10.1136/injuryprev-2019-043286. Epub 2020 Jan 15. PMID 31941758
- [Result] Kwan MM, Close JC, Wong AK, Lord SR. Falls incidence, risk factors, and consequences in Chinese older people: a systematic review. J Am Geriatr Soc. 2011 Mar;59(3):536-43. doi: 10.1111/j.1532-5415.2010.03286.x. Epub 2011 Mar 1. PMID 21361880
- [Result] Schwartz AV, Sellmeyer DE, Ensrud KE, Cauley JA, Tabor HK, Schreiner PJ, Jamal SA, Black DM, Cummings SR; Study of Osteoporotic Features Research Group. Older women with diabetes have an increased risk of fracture: a prospective study. J Clin Endocrinol Metab. 2001 Jan;86(1):32-8. doi: 10.1210/jcem.86.1.7139. PMID 11231974
- [Result] Roman de Mettelinge T, Cambier D, Calders P, Van Den Noortgate N, Delbaere K. Understanding the relationship between type 2 diabetes mellitus and falls in older adults: a prospective cohort study. PLoS One. 2013 Jun 25;8(6):e67055. doi: 10.1371/journal.pone.0067055. Print 2013. PMID 23825617
- [Result] Tilling LM, Darawil K, Britton M. Falls as a complication of diabetes mellitus in older people. J Diabetes Complications. 2006 May-Jun;20(3):158-62. doi: 10.1016/j.jdiacomp.2005.06.004. PMID 16632235
- [Result] Chiba Y, Kimbara Y, Kodera R, Tsuboi Y, Sato K, Tamura Y, Mori S, Ito H, Araki A. Risk factors associated with falls in elderly patients with type 2 diabetes. J Diabetes Complications. 2015 Sep-Oct;29(7):898-902. doi: 10.1016/j.jdiacomp.2015.05.016. Epub 2015 Jun 1. PMID 26122285
- [Result] Johnston SS, Conner C, Aagren M, Ruiz K, Bouchard J. Association between hypoglycaemic events and fall-related fractures in Medicare-covered patients with type 2 diabetes. Diabetes Obes Metab. 2012 Jul;14(7):634-43. doi: 10.1111/j.1463-1326.2012.01583.x. Epub 2012 Mar 14. PMID 22335246
- [Result] Maurer MS, Burcham J, Cheng H. Diabetes mellitus is associated with an increased risk of falls in elderly residents of a long-term care facility. J Gerontol A Biol Sci Med Sci. 2005 Sep;60(9):1157-62. doi: 10.1093/gerona/60.9.1157. PMID 16183956
- [Result] Albornos-Munoz L, Moreno-Casbas MT, Sanchez-Pablo C, Bays-Moneo A, Fernandez-Dominguez JC, Rich-Ruiz M, Gea-Sanchez M; Otago Project Working Group. Efficacy of the Otago Exercise Programme to reduce falls in community-dwelling adults aged 65-80 years old when delivered as group or individual training. J Adv Nurs. 2018 Jul;74(7):1700-1711. doi: 10.1111/jan.13583. Epub 2018 Jun 3. PMID 29633328
- [Result] Sinclair A, Saeedi P, Kaundal A, Karuranga S, Malanda B, Williams R. Diabetes and global ageing among 65-99-year-old adults: Findings from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2020 Apr;162:108078. doi: 10.1016/j.diabres.2020.108078. Epub 2020 Feb 14. PMID 32068097
- [Result] Salari N, Darvishi N, Ahmadipanah M, Shohaimi S, Mohammadi M. Global prevalence of falls in the older adults: a comprehensive systematic review and meta-analysis. J Orthop Surg Res. 2022 Jun 28;17(1):334. doi: 10.1186/s13018-022-03222-1. PMID 35765037
- [Result] Barrett-Connor E, Weiss TW, McHorney CA, Miller PD, Siris ES. Predictors of falls among postmenopausal women: results from the National Osteoporosis Risk Assessment (NORA). Osteoporos Int. 2009 May;20(5):715-22. doi: 10.1007/s00198-008-0748-2. Epub 2008 Sep 17. PMID 18797811
- [Result] Gale CR, Cooper C, Aihie Sayer A. Prevalence and risk factors for falls in older men and women: The English Longitudinal Study of Ageing. Age Ageing. 2016 Nov;45(6):789-794. doi: 10.1093/ageing/afw129. Epub 2016 Jul 19. PMID 27496938
- [Result] Zia A, Kamaruzzaman SB, Tan MP. Polypharmacy and falls in older people: Balancing evidence-based medicine against falls risk. Postgrad Med. 2015 Apr;127(3):330-7. doi: 10.1080/00325481.2014.996112. Epub 2014 Dec 24. PMID 25539567
- [Result] Tinetti ME, Williams CS. The effect of falls and fall injuries on functioning in community-dwelling older persons. J Gerontol A Biol Sci Med Sci. 1998 Mar;53(2):M112-9. doi: 10.1093/gerona/53a.2.m112. PMID 9520917
- [Result] Friedman SM, Munoz B, West SK, Rubin GS, Fried LP. Falls and fear of falling: which comes first? A longitudinal prediction model suggests strategies for primary and secondary prevention. J Am Geriatr Soc. 2002 Aug;50(8):1329-35. doi: 10.1046/j.1532-5415.2002.50352.x. PMID 12164987
- [Result] Demura S, Yamada T, Kasuga K. Severity of injuries associated with falls in the community dwelling elderly are not affected by fall characteristics and physical function level. Arch Gerontol Geriatr. 2012 Jul-Aug;55(1):186-9. doi: 10.1016/j.archger.2011.06.033. Epub 2011 Jul 27. PMID 21794930
- [Result] Alexander BH, Rivara FP, Wolf ME. The cost and frequency of hospitalization for fall-related injuries in older adults. Am J Public Health. 1992 Jul;82(7):1020-3. doi: 10.2105/ajph.82.7.1020. PMID 1609903
- [Result] Burns ER, Lee R, Hodge SE, Pineau VJ, Welch B, Zhu M. Validation and comparison of fall screening tools for predicting future falls among older adults. Arch Gerontol Geriatr. 2022 Jul-Aug;101:104713. doi: 10.1016/j.archger.2022.104713. Epub 2022 Apr 30. PMID 35526339
- [Result] Park SH, Lee YS. The Diagnostic Accuracy of the Berg Balance Scale in Predicting Falls. West J Nurs Res. 2017 Nov;39(11):1502-1525. doi: 10.1177/0193945916670894. Epub 2016 Oct 26. PMID 27784833
- [Result] Vongsirinavarat M, Mathiyakom W, Kraiwong R, Hiengkaew V. Fear of Falling, Lower Extremity Strength, and Physical and Balance Performance in Older Adults with Diabetes Mellitus. J Diabetes Res. 2020 Jun 3;2020:8573817. doi: 10.1155/2020/8573817. eCollection 2020. PMID 32587870
- [Result] Pijpers E, Ferreira I, de Jongh RT, Deeg DJ, Lips P, Stehouwer CD, Nieuwenhuijzen Kruseman AC. Older individuals with diabetes have an increased risk of recurrent falls: analysis of potential mediating factors: the Longitudinal Ageing Study Amsterdam. Age Ageing. 2012 May;41(3):358-65. doi: 10.1093/ageing/afr145. Epub 2011 Dec 8. PMID 22156559
- [Result] Panel on Prevention of Falls in Older Persons, American Geriatrics Society and British Geriatrics Society. Summary of the Updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011 Jan;59(1):148-57. doi: 10.1111/j.1532-5415.2010.03234.x. PMID 21226685
- [Result] Ligthelm RJ, Kaiser M, Vora J, Yale JF. Insulin use in elderly adults: risk of hypoglycemia and strategies for care. J Am Geriatr Soc. 2012 Aug;60(8):1564-70. doi: 10.1111/j.1532-5415.2012.04055.x. Epub 2012 Aug 6. PMID 22881394
- [Result] Yau RK, Strotmeyer ES, Resnick HE, Sellmeyer DE, Feingold KR, Cauley JA, Vittinghoff E, De Rekeneire N, Harris TB, Nevitt MC, Cummings SR, Shorr RI, Schwartz AV. Diabetes and risk of hospitalized fall injury among older adults. Diabetes Care. 2013 Dec;36(12):3985-91. doi: 10.2337/dc13-0429. Epub 2013 Oct 15. PMID 24130352
- [Result] Berlie HD, Garwood CL. Diabetes medications related to an increased risk of falls and fall-related morbidity in the elderly. Ann Pharmacother. 2010 Apr;44(4):712-7. doi: 10.1345/aph.1M551. Epub 2010 Mar 9. PMID 20215495
- [Result] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Result] Sherrington C, Fairhall N, Kwok W, Wallbank G, Tiedemann A, Michaleff ZA, Ng CACM, Bauman A. Evidence on physical activity and falls prevention for people aged 65+ years: systematic review to inform the WHO guidelines on physical activity and sedentary behaviour. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):144. doi: 10.1186/s12966-020-01041-3. PMID 33239019
- [Result] Thomas S, Mackintosh S, Halbert J. Does the 'Otago exercise programme' reduce mortality and falls in older adults?: a systematic review and meta-analysis. Age Ageing. 2010 Nov;39(6):681-7. doi: 10.1093/ageing/afq102. Epub 2010 Sep 4. PMID 20817938
- [Result] Martins AC, Santos C, Silva C, Baltazar D, Moreira J, Tavares N. Does modified Otago Exercise Program improves balance in older people? A systematic review. Prev Med Rep. 2018 Jul 10;11:231-239. doi: 10.1016/j.pmedr.2018.06.015. eCollection 2018 Sep. PMID 30210995
- [Result] Chapman A, Meyer C, Renehan E, Hill KD, Browning CJ. Exercise interventions for the improvement of falls-related outcomes among older adults with diabetes mellitus: A systematic review and meta-analyses. J Diabetes Complications. 2017 Mar;31(3):631-645. doi: 10.1016/j.jdiacomp.2016.09.015. Epub 2016 Sep 30. PMID 27765575
- [Result] Shier V, Trieu E, Ganz DA. Implementing exercise programs to prevent falls: systematic descriptive review. Inj Epidemiol. 2016 Dec;3(1):16. doi: 10.1186/s40621-016-0081-8. Epub 2016 Jul 4. PMID 27747553
- [Result] Teng B, Gomersall SR, Hatton A, Brauer SG. Combined group and home exercise programmes in community-dwelling falls-risk older adults: Systematic review and meta-analysis. Physiother Res Int. 2020 Jul;25(3):e1839. doi: 10.1002/pri.1839. Epub 2020 May 11. PMID 32394595
- [Result] Thanapluetiwong S, Chewcharat A, Takkavatakarn K, Praditpornsilpa K, Eiam-Ong S, Susantitaphong P. Vitamin D supplement on prevention of fall and fracture: A Meta-analysis of Randomized Controlled Trials. Medicine (Baltimore). 2020 Aug 21;99(34):e21506. doi: 10.1097/MD.0000000000021506. PMID 32846760
- [Result] Bischoff-Ferrari HA, Dawson-Hughes B, Staehelin HB, Orav JE, Stuck AE, Theiler R, Wong JB, Egli A, Kiel DP, Henschkowski J. Fall prevention with supplemental and active forms of vitamin D: a meta-analysis of randomised controlled trials. BMJ. 2009 Oct 1;339:b3692. doi: 10.1136/bmj.b3692. PMID 19797342
- [Result] Montero-Odasso M, van der Velde N, Martin FC, Petrovic M, Tan MP, Ryg J, Aguilar-Navarro S, Alexander NB, Becker C, Blain H, Bourke R, Cameron ID, Camicioli R, Clemson L, Close J, Delbaere K, Duan L, Duque G, Dyer SM, Freiberger E, Ganz DA, Gomez F, Hausdorff JM, Hogan DB, Hunter SMW, Jauregui JR, Kamkar N, Kenny RA, Lamb SE, Latham NK, Lipsitz LA, Liu-Ambrose T, Logan P, Lord SR, Mallet L, Marsh D, Milisen K, Moctezuma-Gallegos R, Morris ME, Nieuwboer A, Perracini MR, Pieruccini-Faria F, Pighills A, Said C, Sejdic E, Sherrington C, Skelton DA, Dsouza S, Speechley M, Stark S, Todd C, Troen BR, van der Cammen T, Verghese J, Vlaeyen E, Watt JA, Masud T; Task Force on Global Guidelines for Falls in Older Adults. World guidelines for falls prevention and management for older adults: a global initiative. Age Ageing. 2022 Sep 2;51(9):afac205. doi: 10.1093/ageing/afac205. PMID 36178003
- See also: United Nations Department of Economic and Social Affairs, Population Division. World Population Ageing 2020 Highlights — https://www.un.org/development/desa/pd/news/world-population-ageing-2020-highlights

DOCUMENTS (1):
  • Informed Consent Form (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT06345118/ICF_000.pdf